CLINICAL TRIAL: NCT02392741
Title: Effects of a Physical Exercise Program on Microcirculation and Pregnancy Outcomes in Obese Pregnant Women: Randomized Clinical Trial
Brief Title: Effects of a Physical Exercise Program on Microcirculation and Pregnancy Outcomes in Obese Pregnant Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Karine Ferreira Agra (Other)
Collaborators: Professor Fernando Figueira Integral Medicine Institute (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor-Investigator, Karine Ferreira Agra, Master in Health, Professor Fernando Figueira Integral Medicine Institute
Organization: Professor Fernando Figueira Integral Medicine Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1161-5873
Record Dates: First submitted 2015-02-25; First posted 2015-03-19 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Obesity; Pregnancy
Keywords: Physical Activity; Microcirculation; Pregnancy Outcome; Obesity; Pregnancy
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): The control group will follow the IMIP prenatal routine.
- Physical exercise program (Experimental): The intervention group witch will be submitted to an exercise program consisting of daily post prandial, 10' after breakfast, lunch and dinner.
  Interventions: Other: Physical exercise program

INTERVENTIONS:
Other: Physical exercise program — The intervention consists to an exercise program composed by a daily post prandial, 10' after breakfast, lunch and dinner, totaling 150' weekly, for eight weeks.
  Other Names: Walking
  Arms: Physical exercise program

SUMMARY:
This study aims to determine the effect of a physical exercise program on microcirculation and maternal and perinatal outcomes in obese women. A randomized clinical trial will be performed at IMIP with obese pregnant women assisted at the Instituto de Medicina Integral Professor Fernando Figueira (IMIP) prenatal service.

DETAILED DESCRIPTION:
Obesity in pregnancy is an important risk factor for adverse perinatal outcomes. Obesity leads to oxidative stress and vascular damage including microcirculation inflammation. Physical activity prevents cellular damage and provide a protective effect to the health of the mother and fetus. Although physical activity has been recommended for obese pregnant women, studies assessing the effects on the microcirculation of these women are scarce. This study aims to determine the effect of a physical exercise program on microcirculation and maternal and perinatal outcomes in obese women. A randomized clinical trial will be performed at IMIP with obese pregnant women assisted at the IMIP prenatal service. The intervention group will be submitted to an exercise program consisting of daily post prandial, 10' after breakfast, lunch and dinner. The control group will follow the routine prenatal IMIP. All pregnant women will be evaluated by a questionnaire to assess physical activity. Microcirculation function will be evaluated by a Laser-doppler flowmetry at baseline and eight weeks after intervention. All pregnant women will be followed until the delivery and immediate postpartum period to check their perinatal outcomes. All pregnant women will be advised to use a pedometer to record their daily steps. The study meets the recommendations of the National Health Council. This project was submitted and approved from the Ethics Committee for Research involving human subjets of IMIP. All participants will be duly informed about the aims of the study and will be included after signing the Informed Consent Form.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy between 14 and 20 weeks gestation;
* Literate women;
* sedentary lifestyle.

Exclusion Criteria:

* Cognitive, auditory, visual or motor impairment, certified by a specialist;
* Any pregnancy disorders or previous maternal diseases: diabetes type 1 or type 2, hypertensive disorders of pregnancy, hemodynamic instability, renal disease or collagen, vaginal bleeding;
* Any medical or obstetric contraindication to perform physical activity.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Effects on microcirculation | change from baseline microcirculation after 8 weeks
  Microcirculation will be assessed using the Laser-doppler flowmetry manufacturers software (Moor Instruments, UK) and expressed in perfusion units (PU). The parameters that will be used to evaluate the microcirculation (microvascular function) are: resting skin blood flux (RF), maximum skin blood flux (MF) at peak PORH, the ratio of maximum level and flow at rest (MF/RF) and the area of hyperemia (AH) which is the graphical area under the curve formed during PORH.

SECONDARY OUTCOMES:
Gestational diabetes | at 30 weeks gestation
  glucose> 92mg / dl before ingestion of 75g of glucose; glucose> 180 mg / dl one hour after the ingestion of 75g of glucose; glucose> 153 mg / dL during the second hour after ingestion of 75 g glucose.
Gestational hypertension | at 30 weeks gestation
  hypertension diagnosed after the twentieth week of gestation in previously normotensive women, which is not accompanied by proteinuria. Nominal and dichotomous variable of yes/no.
Preeclampsia | at 30 weeks gestation
  Hypertension accompanied by proteinuria> 300 mg in a sample of 24 hours (or 1+ in qualitative dipstick test). Nominal and dichotomous variable of yes / no.
Weight gain | at admission on the study and till 40 weeks gestation
  refers to the weight gain (kg) during pregnancy. Obtained from the difference between the weight in late pregnancy and the previous weight before pregnancy - numeric variable, continuous.
Gestational age at delivery | at delivery
  gestational age at delivery measured in complete weeks - numeric variable and discrete
Maternal death | within 42 days of termination of pregnancy
  death of women during or within 42 days of termination of pregnancy, irrespective of the duration or location of the pregnancy, caused by any factor related to or aggravated by pregnancy or by measures taken in relation to it. Nominal variable, dichotomous yes / no.
birth weight | at birth
  quantitative and continuous variable measures in grams.
birth height | at birth
  quantitative and continuous variable measured in centimeters.
Apgar score | at birth
  scale ranging from one to ten according to health conditions at birth. Nominal variable, dichotomous type (one to ten).
head circumference | at birth
  head circumference of newborns measured in centimeters, according to the registration statement of anthropometric characteristics at birth.
Waist circumference | at birth
  waist circumference of the newborn measured in centimeters, according to the registration statement of anthropometric characteristics at birth. Numerical variable, continuous.
Occurrence of birth trauma | at birth
  information obtained through medical records. Nominal variable, dichotomous yes / no.
necessity of hospitalization in the first week of life | one week after delivery
  information obtained through medical records. Nominal variable, dichotomous yes / no.
fetal or neonatal death | after delivery
  information obtained by death certificate. Nominal variable, dichotomous yes / no.

CONTACTS AND LOCATIONS:
Overall Officials: José Roberto da Silva Junior, Master, Study Director — Professor Fernando Figueira Integral Medicine Institute; Isabelle Eunice de Albuquerque Pontes, Master, Study Chair — Professor Fernando Figueira Integral Medicine Institute; João Guilherme Bezerra Alves, PhD, Principal Investigator — Professor Fernando Figueira Integral Medicine Institute; Karine Ferreira Agra, Master, Study Chair — Professor Fernando Figueira Integral Medicine Institute